CLINICAL TRIAL: NCT01444066
Title: The Role Of Empiric Dilation In Patients With Dysphagia With Normal Endoscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201106053
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Dysphagia With Normal Endoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dilation to 27 French (Placebo Comparator)
  Interventions: Procedure: Dilation of the esophagus
- Dilation of the esophagus to 54 French (Experimental): Esophagus will be dilated with a Savory dilator
  Interventions: Procedure: Dilation of the esophagus

INTERVENTIONS:
Procedure: Dilation of the esophagus — Esophagus will be dilated with a Savory dilator.

SUMMARY:
The goal of our study is to determine if stretching the esophagus with a rubber dilator helps patients with swallowing difficulties who have a normal appearing esophagus on upper endoscopy. In order to do this we will perform a randomized controlled study, where patients will undergo esophageal dilation (stretching) with different diameter dilators. We will measure change in symptom severity between baseline (prior to dilation) and 1, 3, 6 and 12 months after the procedure

DETAILED DESCRIPTION:
Dysphagia typically refers to the sensation of food being stuck in the throat or chest( esophageal dysphagia) as well as difficulty with the initiation of swallowing (oropharyngeal dysphagia). It is typically classified into oropharyngeal and esophageal dysphagia. Oropharyngeal dysphagia is typically the result of neuromuscular disease as well as head and neck malignancy and can be diagnosed on the basis of history and physical examination in most cases. Patients with esophageal dysphagia can further be sub-classified into two groups; those with obvious abnormality in the esophageal mucosa or motility on endoscopy and those with normal findings on endoscopic examination.

The diagnosis and treatment of patients with dysphagia and abnormal findings on endoscopy has been extensively studied and there are well-define practice guidelines availed on the subject. In contrast to this the management strategy for the group of patients with esophageal type dysphagia and a normal appearing esophagus on upper endoscopy (DNE) has been a topic of controversy for over a decade. Those patients with DNE are thought to fall into several categories, those with very subtle strictures and rings in the esophagus that are not seen during endoscopy, as well as patients with non-erosive reflux disease, eosinophilic esophagitis, primary motility disorders of the esophagus, and finally those with "functional" dysphagia (in whom no cause can be identified). Several approaches have been advocated for the evaluation and treatment of patients with DNE, including a trial of proton pump inhibitor therapy, obtaining random biopsies to exclude eosinophilic esophagitis and non-erosive reflux disease, referral for manometry and esophageal pH monitoring, as well as empiric esophageal dilation with a large caliber bougie. Of these options empiric esophageal dilation with a large diameter bougie has been the initial management approach recommended by the most recent AGA guidelines as well as many experts in the field of esophagology, for the treatment of DNE.

The initial evidence for empiric esophageal dilation in patients with DNE came from a retrospective study by Marshal et al, who found that 50% of patients experienced a sustained improvement in symptoms following dilation with a large diameter bougie. This was followed by a randomized controlled trial by Colon and coworkers, who again found a significant benefit to empiric esophageal bougie dilation. However, two randomized trials in the mid-2000's did not find any benefit to empiric esophageal dilation; although the dilation methods used in these studies differed from that used by Marshal and Colon et al. Despite these conflicting results empiric dilation continues to be popular by community gastroenterologists, and is perceived to be safe effective intervention for treating patients with DEN. A recent study by Olson et al found that empiric dilation for DNE was performed more commonly then dilation for dilation for esophageal strictures in the United States and is associated with a 0.65% complication rate. Additionally, in the current era of financial pressure on the medical community empiric dilation for DNE at the time of the first diagnostic upper endoscopy could lead to a significant savings if it is effective in relieving symptoms; by obviating the need for further diagnostic testing, medications and repeat endoscopy.

With this in mind, our goal is to conduct a randomized controlled trial evaluating the role of empiric dilation in patients with DNE, to help fill existing gaps in the medical literature. Specifically, prior studies are lacking with regard to three important points. First, esophageal manometry and pH monitoring were not uniformly performed on patients; this testing is crucial to excluding esophageal motility disorders and non-erosive reflux disease, which are thought to be causes of DNE. Second, esophageal biopsies were not performed in any of the studies; this has become a standard part of the evaluation of all patients with DNE over the past 5 years, as eosinophilic esophagitis and non-erosive reflux disease can lead to dysphagia and may be missed without microscopic examination of the esophageal mucosa. Finally, none of the studies used a standardized and validated dysphagia questionnaire, such as the Mayo Dysphagia Questionnaire (MDQ) to evaluate symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age: > 18 years.
2. Outpatients undergoing EGD for dysphagia.
3. Ability to provide written informed consent.

Exclusion Criteria:

* Abnormal endoscopy (stricture, abnormal motility or mucosa observed)
* Oropharyngeal dysphagia suspected based on history and physical examination
* History of CVA or other neurologic disorder
* Known connective tissue disease (SLE, scleroderma, CREST, RA)
* Known histopathology based esophageal motor disorder, e.g. achalasia
* Prior thoracic or foregut surgery (excluding cholecystectomy)
* Prior thoracic radiation therapy
* Hiatus hernia >2 cm as judged during EGD

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2013-10-24 (Actual); Study Completion 2013-10-24 (Actual)

PRIMARY OUTCOMES:
Improvement in dysphagia, quantified using 10 cm VAS scale | 12 months

SECONDARY OUTCOMES:
Evaluate the yield of esophageal biopsy in patients with dysphagia with normal endoscopy | 12 months
Evaluate the yield of HRM and pH monitoring in patients with dysphagia and normal endoscopy | 12 months
Identify predictors of response to empiric dilation in patients with dysphagia and normal endoscopy | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Barnes Jewish Hospital, St Louis, Missouri
  - Washington University, St Louis, Missouri